CLINICAL TRIAL: NCT01475643
Title: Safety and Efficacy of Topical Loteprednol Etabonate 0.5%, Versus Prednisolone Acetate 1%, for the Treatment of Intraocular Inflammation Following Surgery for Childhood Cataract
Brief Title: Loteprednol vs Prednisolone for the Treatment of Intraocular Inflammation Following Cataract Surgery in Children.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 670
Record Dates: First submitted 2011-11-17; First posted 2011-11-21 (Estimated); Results first posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Cataract
Keywords: Pediatric cataract
MeSH Terms: conditions — Cataract | interventions — Loteprednol Etabonate

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Loteprednol etabonate (Experimental): Loteprednol etabonate 0.5%
  Interventions: Drug: Loteprednol etabonate
- Prednisolones acetate (Active Comparator): Prednisolone acetate 1.0%
  Interventions: Drug: Prednisolones acetate

INTERVENTIONS:
Drug: Loteprednol etabonate — 1-2 Ophthalmic drops administered to study eye four times daily (QID) for 14 days post surgery. Tapered to twice daily (BID) for 7 days. Then once daily (QD) for 7 days.
  Other Names: LE
  Arms: Loteprednol etabonate
Drug: Prednisolones acetate — 1-2 Ophthalmic drops administered to study eye four times daily (QID) for 14 days post surgery. Tapered to twice daily (BID) for 7 days. Then once daily (QD) for 7 days.
  Other Names: PA
  Arms: Prednisolones acetate

SUMMARY:
The objective of this study is to compare the efficacy and safety for the treatment of postoperative inflammation following ocular surgery for childhood cataract.

DETAILED DESCRIPTION:
The objective of this study is to compare the efficacy and safety of topical Loteprednol Etabonate (LE), 0.5%, to Prednisolone Acetate 1%, for the treatment of postoperative inflammation following ocular surgery for childhood cataract.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a candidate for routine, uncomplicated surgery for childhood cataract

Exclusion Criteria:

* Subjects who have a severe/serious ocular condition, or any other unstable medical condition that, in the Investigator's opinion, may preclude study treatment or follow-up.
* Subjects with glaucoma, ocular hypertension, or those receiving intraocular pressure (IOP) lowering therapy in either eye or systemically.
* Subjects with a history of steroid-induced IOP elevation in either eye.
* Subjects who have known hypersensitivity or other contraindication to the study drug(s) or any components in the drug formulation.

Max Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 107 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson Varughese, Study Director — Valeant/Bausch & Lomb
Locations (1):
- Bausch & Lomb Inc, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Loteprednol Etabonate | Prednisolones Acetate
Started | 54 (53 included in Intent-to-treat (ITT) population, due to no post-treatment assessment.) | 53 (52 included in Intent-to-treat (ITT) population, due to no post-treatment assessment.)
Completed | 40 | 43
Not Completed | 14 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Loteprednol Etabonate | Prednisolones Acetate | Total
Number analyzed (Participants) | 53 | 52 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.7 (3.22) | 4.3 (3.39) | 4 (3.305)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 26 | 48
  Male | 31 | 26 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 20 | 44
  Not Hispanic or Latino | 29 | 32 | 61
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 18 | 18 | 36
  Black or African American | 8 | 10 | 18
  White | 26 | 23 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 53 | 52 | 105

OUTCOME MEASURES:

1. Primary Outcome: Anterior Chamber Inflammation
Description: Anterior Chamber Inflammation (for subjects that could only be examined with a pen light and a 20D [g20 Diopter] magnifying lens): 0 = None Clear anterior chamber with no visible clouding (Tyndall effect and cells combined). Red reflex normal
  1. = Mild Mild anterior chamber clouding. Clear iris pattern on visualization. Red reflex normal
  2. = Moderate Moderate anterior chamber clouding
  3. = Severe Severe anterior chamber clouding. Iris pattern not clearly visualized. Red reflex diminished
  4. = Very severe Severe anterior chamber clouding with a white and/or milky appearance of the anterior chamber. Red reflex absent or severely diminished
Time Frame: Postoperative Day 29
Population: Proportion of subjects with anterior chamber inflammation
Measure: Mean (95% Confidence Interval); unit: grade of anterior chamber cells
Arm/Group | Loteprednol Etabonate | Prednisolones Acetate
Number analyzed (Participants) | 53 | 48
grade of anterior chamber cells | .913 [.668 to 1.158] | .783 [.528 to 1.038]

2. Secondary Outcome: Anterior Chamber Cells & Flare
Description: Anterior Chamber Flare (for those subjects that could be examined with a slit lamp):
  Assessed scattering of a slit lamp light beam when directed into the anterior chamber (Tyndall effect). 0 = None No Tyndall effect
  1. = Mild Tyndall effect barely discernible
  2. = Moderate Tyndall effect in anterior chamber is moderately intense. Iris pattern is seen clearly
  3. = Severe Tyndall effect in anterior chamber is severely intense. Iris pattern cannot be seen clearly
  4. = Very severe Tyndall effect is very severely intense. The aqueous has a white and milky appearance
Time Frame: Over all visits 42 days
Population: Proportion of subjects with anterior chamber flare.
Measure: Mean (95% Confidence Interval); unit: Grade of anterior chamber flare
Arm/Group | Loteprednol Etabonate | Prednisolones Acetate
Number analyzed (Participants) | 36 | 42
Grade of anterior chamber flare | .192 [.034 to .350] | .341 [.157 to .507]

ADVERSE EVENTS:
Time Frame: 29 days
Description: The period of observation for collection of Adverse Events (AEs) extended from the time the subject's parent/legal guardian gave informed consent until the last study visit, Visit 8 (Postoperative Day 90).
Arm/Group | Loteprednol Etabonate | Prednisolones Acetate
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/53
Serious Adverse Events (participants affected / at risk) | 3/54 | 0/53
Other Adverse Events (participants affected / at risk) | 34/54 | 23/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Loteprednol Etabonate (N=54) | Prednisolones Acetate (N=53)
Vitreous Disorder (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 2 (2) | 0 (0)
Bronchiolitis (Eye disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Loteprednol Etabonate (N=54) | Prednisolones Acetate (N=53)
Amblyopia (Eye disorders) | 1 (1) | 1 (1)
cataract (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Eye Pain (Eye disorders) | 6 (6) | 4 (4)
Eyelid Odema (Eye disorders) | 4 (4) | 4 (4)
Glaucoma (Eye disorders) | 2 (4) | 0 (0)
Ocular hyperemia (Eye disorders) | 3 (3) | 0 (0)
Iridocyclitis (Eye disorders) | 0 (0) | 1 (1)
lacrimation increased (Eye disorders) | 1 (1) | 0 (0)
Strabismus (Eye disorders) | 1 (1) | 0 (0)
Vitreous Disorder (Eye disorders) | 1 (1) | 0 (0)
photophobia (Eye disorders) | 1 (1) | 0 (0)
Suture Related Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Discomfort (General disorders) | 2 (2) | 3 (3)
Installation Site Pain (General disorders) | 0 (0) | 1 (1)
injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Post Procedural Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post Capsule Opacification (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
iritis (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Feeling Hot (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Ear Infection (Infections and infestations) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (3) | 4 (4)
Gastroenteritis Viral (Infections and infestations) | 2 (2) | 1 (1)
Pharyngitis Strepococcal (Infections and infestations) | 1 (1) | 0 (0)
Arthropod Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2013-05-22): https://cdn.clinicaltrials.gov/large-docs/43/NCT01475643/Prot_000.pdf
  • Statistical Analysis Plan (2013-05-22): https://cdn.clinicaltrials.gov/large-docs/43/NCT01475643/SAP_001.pdf